CLINICAL TRIAL: NCT07275723
Title: A Multicenter, Randomized, Double-Blind, Positive-Controlled, Cross-Over Phase III Clinical Trial Evaluating the Efficacy and Safety of HRS-9231 for Body Parts (Non-Central Nervous System) Magnetic Resonance Imaging (MRI)
Brief Title: A Study of a Gadolinium-Based Contrast Agent (GBCA) for Adults Undergoing Magnetic Resonance Imaging (MRI) for Known or Highly Suspected Body Parts (Non-Central Nervous System) Lesions
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Shengdi Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: HRS-9231-302
Record Dates: First submitted 2025-11-18; First posted 2025-12-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: For Contrast-enhanced Magnetic Resonance Imaging (MRI) of Abnormal Vascular Lesions in Body Regions Excluding the Central Nervous System (CNS)
MeSH Terms: interventions — gadobutrol; Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-9231 + Gadobutrol Group (Experimental): HRS-9231 enhanced MRI then Gadobutrol enhanced MRI.
  Interventions: Drug: HRS-9231 Injection; Drug: Gadobutrol Injection; Device: Magnetic Resonance Imaging (MRI)
- Gadobutrol + HRS-9231 Group (Experimental): Gadobutrol enhanced MRI then HRS-9231 enhanced MRI.
  Interventions: Drug: HRS-9231 Injection; Drug: Gadobutrol Injection; Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Drug: HRS-9231 Injection — HRS-9231 injection.
Drug: Gadobutrol Injection — Gadobutrol injection.
Device: Magnetic Resonance Imaging (MRI) — Magnetic Resonance Imaging (MRI).

SUMMARY:
The purpose of this study is to evaluate the efficacy of HRS-9231 for Magnetic Resonance Imaging (MRI) of body regions excluding the Central Nervous System (CNS) in patients undergoing MRI examinations, using the patient's own unenhanced MRI images as a control; to demonstrate that the efficacy of HRS-9231 is not inferior to gadobutrol for lesion visualization in body MRI; to evaluate the safety of HRS-9231 for body MRI; and to explore the population pharmacokinetic characteristics of HRS-9231 in subjects undergoing body MRI examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent, be willing and able to comply with study requirements.
2. Age ≥18 years, male or female.
3. Subjects who are scheduled to undergo a contrast-enhanced MRI (including MRA) examination and who, within 12 months prior to signing the informed consent form, have had imaging examinations that identified at least one known or highly suspected region of enhancement abnormality or lesion in the body.

Exclusion Criteria:

1. Investigator judges unstable clinical condition or comorbidities that may affect MRI image comparability or study parameters.
2. Severe renal impairment (baseline eGFR < 30 mL/min/1.73m²) before first dose; acute kidney injury regardless of eGFR.
3. Acute kidney injury, irrespective of eGFR levels.
4. Contraindication to MRI or gadolinium contrast agents.
5. History of severe allergic reactions to drugs, contrast agents, or other allergens.
6. Severe cardiovascular disease.
7. Pregnant or breastfeeding women.
8. Any other condition deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
To compare the lesion visualization scores (border delineation) of HRS-9231-enhanced with gadobutrol-enhanced MRI. | Day 1 after procedure.
To compare the lesion visualization scores (internal morphology) of HRS-9231-enhanced with gadobutrol-enhanced MRI. | Day 1 after procedure.
To compare the lesion visualization scores (degree of contrast enhancement) of HRS-9231-enhanced with gadobutrol-enhanced MRI. | Day 1 after procedure.

SECONDARY OUTCOMES:
To compare the lesion visualization scores of HRS-9231-enhanced with unenhanced MRI. | Day 1 after procedure.
Number and size of lesions in MRI images after receiving HRS-9231. | Day 1 after procedure.
Number and size of lesions in MRI images after receiving the control drug. | Day 1 after procedure.
HRS-9231 plasma concentration. | Day 1 after procedure.
Population pharmacokinetic parameters - clearance. | Day 1 after procedure.
Population pharmacokinetic parameters - apparent volume of distribution. | Day 1 after procedure.
Sensitivity for lesion detection on MRI images obtained with HRS-9231. | Day 1 after procedure.
Specificity for lesion detection on MRI images obtained with HRS-9231. | Day 1 after procedure.
Sensitivity for lesion detection on MRI images obtained with gadobutrol. | Day 1 after procedure.
Specificity for lesion detection on MRI images obtained with gadobutrol. | Day 1 after procedure.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided